CLINICAL TRIAL: NCT06647095
Title: Identification of New Non-invasive Biomarkers of Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) in Patients by Blood Plasma Spectroscopy, Breath Volatile Organic Compounds Analysis and Serum Bile Acids Analysis
Brief Title: New Non-invasive Biomarkers of Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD)
Status: Completed | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Barbora Nováková, MD, Principal Investigator, General University Hospital, Prague
Other Study IDs: GUHPrague83/21
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Simple Steatosis (SS); Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD); Metabolic Dysfunction-associated Steatohepatitis (MASH)
Keywords: Liver steatosis; Liver fibrosis; MASLD; MASH; Blood spectroscopy; Breath tests; d-Limonene; SYFT-MS; Bile acids; metabolic dysfunction-associated steatotic liver disease; metabolic dysfunction-associated steatohepatitis
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples, exhaled breath samples, urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy controls
  Interventions: Dietary Supplement: D-Limonene Gelcaps; Dietary Supplement: Fish Oil Concentrate, 1000 Mg Oral Capsule
- MASH
  Interventions: Dietary Supplement: D-Limonene Gelcaps; Dietary Supplement: Fish Oil Concentrate, 1000 Mg Oral Capsule
- Steatosis
  Interventions: Dietary Supplement: D-Limonene Gelcaps; Dietary Supplement: Fish Oil Concentrate, 1000 Mg Oral Capsule

INTERVENTIONS:
Dietary Supplement: D-Limonene Gelcaps — Capsules containing d-Limonene will be optionally given during the breath test to all participants of all groups
Dietary Supplement: Fish Oil Concentrate, 1000 Mg Oral Capsule — Capsules containing fish oil will be optionally given during the breath test to all participants of all groups

SUMMARY:
The goal of this observational study is to learn if some components of blood or exhaled breath can diagnose people having more fat in their livers than is normal, because of their poorer metabolic health (for example, because of obesity and diabetes). The main questions it aims to answer are:

1. Can a method find participants with higher liver fat than healthy participants?
2. Can a method find participants in whom higher liver fat was a cause of liver inflammation or stiffness?

Participants will:

* fast overnight
* have a routine blood draw
* easily exhale a few times into a special device or a plastic bag and fill in a short dietary questionnaire (if participating in a breath test)
* optionally swallow capsules with an orange peel extract and fish oil before exhaling, which can help get better results from breath (capsules will be medically safe and approved)

DETAILED DESCRIPTION:
Patients with MASLD and healthy volunteers will be offered an observational study evaluating the diagnostic role of new non-invasive experimental methods (serum bile acids, breath VOC, and plasmatic spectroscopic patterns) assessing the presence and severity of liver fibrosis and steatosis.

First, this study aims to differentiate patients with metabolic dysfunction-associated steatotic liver disease (MASLD) and metabolic dysfunction-associated steatohepatitis (MASH) from healthy controls (or simple steatosis) using three experimental methods.

Second, the investigators aim to stratify patients with MASLD according to the presence/grade of steatosis and fibrosis (any, significant F2-3, advanced F3, cirrhosis F4) using the same methods.

Experimental methods tested in this study include:

1. analyzing the fasting spectrum of serum bile acids using liquid chromatography-mass spectrometry
2. analyzing the disease-specific spectroscopy patterns given by vibrational and chiroptical spectroscopy of blood plasma
3. analyzing trace concentrations of volatile organic compounds (VOC) in exhaled human breath using the Selected ion flow tube mass spectrometry. This contains the so-called stress test to monitor breath VOC (d-Limonene and triethylamine) after their regulated ingestion in the form of capsules

These parameters may eventually be combined with anthropometric and laboratory parameters (such as age or BMI).

Clinical examinations, blood sampling, ultrasound examinations of the liver, and liver elastography will be performed as part of routine care.

The results of the blood parameters can be retrospectively evaluated.

Approximately 60-80 participants in total were anticipated for each method. For patients who participate in breath tests, adequate insurance must be guaranteed.

Statistical processing: individual parameters will be evaluated in an exploratory and a validation group or by the PLS-DA algorithm with repeated cross-validation. A difference of p <0.05 will be considered a statistically significant change.

ELIGIBILITY:
Inclusion Criteria for Participants with MASLD:

* Presence of liver steatosis (detected either by hepatic ultrasonography/CAP/histologically) or MASH/simple steatosis confirmed by liver biopsy
* Absence of secondary causes of fat accumulation in the liver and other liver disease: ruled out other etiologies of liver disease, such as viral hepatitis, drug-induced liver disease, autoimmune liver disease, biliary tract disease, and hereditary metabolic diseases

Inclusion Criteria for Negative Controls:

* Absence of liver disease
* For breath analysis: absence of liver steatosis (normal liver ultrasound image and CAP less than 248 dB/m)
* For plasma spectroscopy and bile acid analysis: Body Mass Index ≤ 25 and waist-hip ratio ≤ 0.95 plus normal liver ultrasound
* Absence of diabetes mellitus and metabolic syndrome
* Normal liver function tests, lipid spectrum, fasting glycemia
* Alcohol intake less than 20 g/ day (women) or 30 g/ day (men)

Exclusion Criteria:

* Non-compliance with the investigation program
* Failure to sign the informed consent form
* Liver biopsy/clinic discrepancy
* For LMN a TMA "stress test": fish, see fruit and citrus fruit allergy
* Pregnancy
* For bile acid analysis: Treatment with BA or BA sequestrants
* For bile acid analysis: Portal hypertension (does not apply for MASH patients)
* For bile acid analysis: Cirrhosis (does not apply for MASH patients)
* For plasma spectroscopy: Cirrhosis
* Anamnesis of alcohol abuse (based on GGT, carbohydrate-deficient transferrin, urinary ethyl-glucuronide, and patient's history)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with MASLD of primary care clinic, healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Serum bile acids concentrations in the MASH/ Steatosis/ Healthy controls | A single day during within the data collection period = between September 2021 and September 2024
  Individual bile acid concentrations in blood serum accessed by LC-MS/MS, measured in µmol/L or expressed as detectable or undetectable
The effect of serum bile acids in the MASH/ Steatosis/ Healthy controls discrimination | A single day during within the data collection period = between September 2021 to September 2024
  To access the effect of serum bile acid concentrations on intergroup discrimination in a discriminant model as measured by model parameters and ROC
Native breath concentrations of volatile organic compounds in the aim groups | Single measurement on one day within 6 weeks (from mid-February 2023 to the end of March 2023)
  Concentrations of VOC in fasting exhaled breath expressed in ppbv
A change in d-Limonene and TMA concentrations before and after the ingestion of capsules containing d-LMN, TMA, ppbv | Baseline, at 150min after capsules ingestion - both on one day within 6 weeks (from mid-February 2023 to the end of March 2023)
  A change in concentration of d-Limonene and TMA in exhaled breath after an overnight fast/ post-ingestion of d-Limonene and TMA-containing capsules, expressed in ppbv
The effect of concentrations of volatile organic compounds in exhaled breath, native and post-ingestion, on the discrimination of the aim groups | On one day within 6 weeks (from mid-February 2023 to the end of March 2023)
  To access the effect of VOC concentrations in exhaled breath, native and after the ingestion of d-Limonene and TMA-containing capsules, on intergroup discrimination in a discriminant model as measured by model parameters and ROC
Peak of d-LMN, and TMA concentration after the ingestion of capsules in the aim groups | At an individually specific time point for each participant that occurs within 4 hours after ingestion of d-Limonene and TMA-containing capsules on a single day within 6 weeks (from mid-February 2023 to the end of March 2023)
  A maximum concentration of d-Limonene and TMA in exhaled breath post-ingestion of d-Limonene and TMA-containing capsules, expressed in ppbv
Spectroscopic patterns of blood plasma | Based on single peripheral blood uptake within the data collection period = between September 2021 and September 2024
  Disease-specific patterns of blood plasma expressed as differences in spectra (their normalized intensity (a.u.)) and regions between the aim groups

CONTACTS AND LOCATIONS:
Overall Officials: Barbora Nováková, MD, Principal Investigator — General University Hospital, Prague
Locations (2):
- Czechia (2):
  - Regional Hospital Liberec, Liberec, Czech Republic
  - General University Hospital in Prague, Prague, Czech Republic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zizalova K, Novakova B, Vecka M, Petrtyl J, Lanska V, Pelinkova K, Smid V, Bruha R, Vitek L, Lenicek M. Serum concentration of taurochenodeoxycholic acid predicts clinically significant portal hypertension. Liver Int. 2023 Apr;43(4):888-895. doi: 10.1111/liv.15481. Epub 2022 Nov 25. PMID 36433660
- [Background] WED-280 Spectroscopy of blood plasma has the potential to differentiate metabolic dysfunction-associated steatohepatitis from steatosis Nováková, Barbora et al. Journal of Hepatology, Volume 80, S539 - S540
- [Background] Puri P, Daita K, Joyce A, Mirshahi F, Santhekadur PK, Cazanave S, Luketic VA, Siddiqui MS, Boyett S, Min HK, Kumar DP, Kohli R, Zhou H, Hylemon PB, Contos MJ, Idowu M, Sanyal AJ. The presence and severity of nonalcoholic steatohepatitis is associated with specific changes in circulating bile acids. Hepatology. 2018 Feb;67(2):534-548. doi: 10.1002/hep.29359. Epub 2017 Dec 23. PMID 28696585
- [Background] Spanel P, Smith D. Quantification of volatile metabolites in exhaled breath by selected ion flow tube mass spectrometry, SIFT-MS. Clin Mass Spectrom. 2020 Feb 13;16:18-24. doi: 10.1016/j.clinms.2020.02.001. eCollection 2020 Apr. PMID 34820516
- [Background] Sinha R, Lockman KA, Homer NZM, Bower E, Brinkman P, Knobel HH, Fallowfield JA, Jaap AJ, Hayes PC, Plevris JN. Volatomic analysis identifies compounds that can stratify non-alcoholic fatty liver disease. JHEP Rep. 2020 Jun 15;2(5):100137. doi: 10.1016/j.jhepr.2020.100137. eCollection 2020 Oct. PMID 32775974
- [Background] Ten-Doménech I, Rienda I, Pérez-Rojas J, et al. Progress and challenges of mid-infrared spectroscopy for liver characterization focusing on steatosis, fibrosis and cancer. Applied Spectroscopy Reviews. 2024;59(4):578-599
- [Background] Targher G, Byrne CD, Tilg H. MASLD: a systemic metabolic disorder with cardiovascular and malignant complications. Gut. 2024 Mar 7;73(4):691-702. doi: 10.1136/gutjnl-2023-330595. PMID 38228377